CLINICAL TRIAL: NCT02672501
Title: Open-labeled, Uncontrolled, Single-arm Pilot Study to Evaluate Cellular Immunotherapy Using CD19-targeted Chimeric Antigen Receptor Engineered T Cells in Patients With Relapsed or Refractory CD19+ B Cell Leukemia
Brief Title: A Study to Assess CD19-targeted Immunotherapy T Cells in Patients With Relapsed or Refractory CD19+ B Cell Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai GeneChem Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Genechem
Record Dates: First submitted 2016-01-25; First posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Leukemia, B-Cell
Keywords: immunotherapy; CAR-T; leukemia
MeSH Terms: conditions — Leukemia, B-Cell; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- anti-CD19-CAR-T cells (Experimental): patients receive chemotherapy(CF, cyclophosphamide and Fludarabine) on day -6 to day -1, then infusied with anti-CD19-CAR-T cells transduced with lentivirus on day 0 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: anti-CD19-CAR-T cells

INTERVENTIONS:
Drug: anti-CD19-CAR-T cells — a 2nd CAR, CD19 as target protein, 4-1BB as co- stimulator, and optimized the spatial conformation by a suitable hinge & transmembrane domain sequences
  Other Names: 2nd CAR-T

SUMMARY:
In the conventional treatment options, B cell leukemia could be treated with chemotherapy drugs or HSCT. But chemotherapy could barely cured leukemia. And HSCT is often limited by lacking of HLA-matched donors, even if those patients who received HSCT still could be relapsed. And now, chimeric antigen receptor modified T cell infusion maybe an effective treatment to solve these problems. The investigators use a 2nd CAR- T with the optimized hinge and transmembrane domain to treat patients with relapsed or refractory B cell leukemia, including relapsed cases after HSCT. The purpose of this study is to assess the safety and efficacy of this 2nd CAR-T cells. At the same time, evaluating the possible and clinical responses of using donor-derived T cells engineered CAR-T cells.

Detailed Description: This study is being conducted to assess anti-CD19-CAR-T cells safety and efficacy in treating patients with B cell leukemia. The investigators constructed a 2nd CAR, CD19 as target protein, 4-1BB as co-stimulator. And optimized the spatial conformation by a suitable hinge & transmembrane domain sequences. The source of T cells for CAR-T is from two aspects, one is autologous, the other is donor-derived (only suitable for patients received HSCT before and relapsed). The infusion dose is (1-5)×106 CAR positive T cells/kg, and the specific cells numbers depend on the situation of individual CAR-T cells preparation.

DETAILED DESCRIPTION:
This study is being conducted to assess anti-CD19-CAR-T cells safety and efficacy in treating patients with B cell leukemia. The investigators constructed a 2nd CAR, using CD19 as target, using 4-1BB as co-stimulator, and optimized the spatial conformation by a suitable hinge and transmembrane domain sequences. The source of T cells used to prepare CAR-T could be either autologous, or donor-derived (only suitable for patients received HSCT before and relapsed). The infusion dose is (1-5)×106 CAR positive T cells/kg, and the specific cells numbers depends on the situation of individual CAR-T cells preparation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CD19+ B-cell leukemia as comfirmed by Flow Cytometry
* Age: 1-70 years old
* Expected survival > 12 weeks
* Creatinine < 2.5 mg/dl
* ALT/AST < 3x normal
* Bilirubin <2.0 mg/dl
* Sucessful test expansion of T-cells
* Adequate venous access for apheresis, and no other contraindications for leukapheresis
* Voluntary informed consent is given

Exclusion Criteria:

* Pregnant or lactating women
* Uncontrolled active infection
* Active hepatitis B or hepatitis C infection
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
* Previously treatment with any gene therapy products
* Feasibility assessment during screening demonstrates<30% transduction of target lymphocytes, or insufficient expansion (<5-fold) in response to CD3/CD28 costimulation
* Active central nervous system leukemia
* Any serious, uncontrolled diseases (including, but not limit to, unstable angina pectoris, congestive heart failure, grade Ш or Ⅳ cardiac disease, serious arrhythmia, liver and kidney disorders or metabolic diseases)

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse event | 6 weeks
  asverse event is evaluated with CTCAE, version 4.0

SECONDARY OUTCOMES:
Number of patients with tumor response | 8 weeks
  summarize tumor response by overal response rates
Detection of transferred T cells in the circulation using quantitative -PCR | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Yang, Doctor, Principal Investigator — Shanghai Changhai Hospital，The Second Military Medical University
Locations (1):
- Shanghai Changhai Hospital，The Second Military Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided